CLINICAL TRIAL: NCT03550404
Title: Improving Native American Elder Access to and Use of Healthcare Through Effective Health System Navigation
Brief Title: Improving Native American Elder Access to and Use of Healthcare
Status: Completed | Type: Observational
Sponsor: Pacific Institute for Research and Evaluation (Other)
Collaborators: University of California, San Diego (Other); University of New Mexico (Other)
Responsible Party: Principal Investigator, Cathleen Willging, Senior Research Scientist/Center Director, Pacific Institute for Research and Evaluation
Other Study IDs: 0784.01.01
Record Dates: First submitted 2018-05-15; First posted 2018-06-08 (Actual); Results first posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Access to Health Care

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Navigators: AIE Navigators will use the Seasons of Care app in the context of their everyday outreach work with AIEs over two four-month intervention periods (P1 and P2). Their goal will be to facilitate health literacy to shift attitudes, beliefs, and behaviors to create a "Culture of Coverage" for AIEs at individual, organizational/community, and policy levels. Separated by distance, the AIE Navigators will receive coaching as necessary, using virtual meeting space, to help refine their implementation skills from a member of the research team with experience in AIE health outreach.
  Interventions: Behavioral: Seasons of Care App
- American Indian Elders (AIEs): Elders will be exposed to the Seasons of Care app when they reach out to navigators for assistance navigating the healthcare system.
  Interventions: Behavioral: Seasons of Care App
- Healthcare providers/staff: This cohort will be exposed to the Seasons of Care app via navigators and their patients.
  Interventions: Behavioral: Seasons of Care App

INTERVENTIONS:
Behavioral: Seasons of Care App — A web-based mobile application (app) called the Seasons of Care Elder Navigation Guide will assist elders, their families/caregivers, healthcare providers, outreach workers, and other community members in navigating healthcare and insurance systems. The app has the added advantage of being easy to update to respond to future changes in health care and insurance, and sustainable because it is not dependent on intensive training, developing, and retaining of individuals in professional navigation positions.

SUMMARY:
This community-driven study features a mixed-method, participatory design to examine help-seeking behavior and healthcare experiences of American Indian elders in New Mexico, in order to develop and evaluate a tailored intervention to enhance knowledge of, access to, and use of insurance and available services to reduce healthcare disparities. This study includes qualitative and quantitative interviews combined with concept mapping and focus groups with American Indian elders and other key stakeholders.

DETAILED DESCRIPTION:
This five-year project was developed by investigators from the Behavioral Health Research Center of the Southwest (BHRCS), a center of the Pacific Institute of Research and Evaluation (PIRE), the Health Committee of the New Mexico Indian Council on Aging (NMICoA), and the University of New Mexico (UNM). The project combines qualitative and quantitative interviews with concept-mapping (CM) techniques and focus groups to study insurance coverage, help-seeking behavior, and the healthcare experiences of American Indian Elders (AIEs) in New Mexico (NM). Practical knowledge grounded in the actual perspectives of AIEs and other key stakeholders may improve healthcare practices and policies for a population largely excluded from national and state discussions of health reform. The study data will also inform the adaptation and development of culturally tailored programming to enrich understanding and facilitate negotiation of a changing landscape of healthcare by AIEs. Our four specific aims are to:

1. Assess how AIEs understand, access, maintain, and use insurance coverage.
2. Characterize AIE help-seeking and healthcare experiences in dominant service delivery settings, i.e., Indian Health Service (IHS), tribally-run 638 facilities, and managed care programs.
3. Identify and compare factors that affect AIE access to health care as perceived by multiple stakeholders, i.e., AIEs, outreach workers (OWs), healthcare staff and providers, public sector administrators, and tribal leaders.
4. Develop and assess implementation feasibility of a structured intervention for OWs that promotes enhanced patient navigation, in addition to healthcare literacy, access, and usage among AIEs.

ELIGIBILITY:
Navigators

Inclusion Criteria:

* Working in a health and health insurance outreach
* Routinely interacting with AIEs as part of their jobs
* Primary service region includes target AIEs.

Exclusion Criteria:

* Not Routinely interacting with AIEs as part of their jobs
* Not willing to be trained in or use the Seasons of Care app

American Indian Elders (AIEs) Inclusion

* Age 55+
* Identifying as AI
* Able to read in English
* Able to consent and complete study procedures
* Interacted with Navigator

Exclusion ● Individuals who cannot read in English or who have not interacted with a pilot test Navigator will not be eligible to participate

Healthcare Staff/providers Inclusion

* Individuals who have been in contact with a pilot test Navigator
* Work in a healthcare facility that serves AIEs in one of our 4 regions

Exclusion

● Individuals who have not interacted with a pilot test Navigator or do not work in a healthcare facility serving our primary population, will not be eligible to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Outreach workers from indigenous communities in the southwest United States, and then the American Indian elders, healthcare staff and providers that interact with those outreach workers.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cathleen Willging, Principal Investigator — Pacific Institute for Research and Evaluation
Locations (1):
- Pacific Institute for Research and Evaluation, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Willging CE, Sommerfeld DH, Jaramillo ET, Lujan E, Bly RS, Debenport EK, Verney SP, Lujan R. "Improving Native American elder access to and use of health care through effective health system navigation". BMC Health Serv Res. 2018 Jun 18;18(1):464. doi: 10.1186/s12913-018-3182-y. PMID 29914446

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We used reputational case selection to identify potential participants who were individuals who provided healthcare navigation services to Elders as part of their everyday work. We approached individuals or administrators at community organizations, healthcare facilities, and tribal agencies with an email or in-person description of the study and an invitation to participate. We followed up at each site with up to three emails, visits, or phone calls.
Pre-assignment Details: Due to the complete closure of tribal communities during the COVID-19 pandemic, zero participants were enrolled and assigned in the "American Indian Elders (AIEs)" and "Healthcare Providers/Staff" Arms/Groups, respectively.
Period: Phase 1
Arm/Group | Navigators | American Indian Elders (AIEs) | Healthcare Providers/Staff
Started | 8 | 0 | 0
Completed | 8 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Phase 2
Arm/Group | Navigators | American Indian Elders (AIEs) | Healthcare Providers/Staff
Started | 8 | 0 | 0
Completed | 4 | 0 | 0
Not Completed | 4 | 0 | 0
Not completed — Unable to complete due to other duties during COVID-19 pandemic | 3 | 0 | 0
Not completed — Vacated position | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Due to complete closure of tribal communities during the COVID-19 pandemic, we were unable to complete baseline measures with any American Indian Elders or healthcare providers/staff
Groups:
- Total: Total of all reporting groups
Arm/Group | Navigators | American Indian Elders (AIEs) | Healthcare Providers/Staff | Total
Number analyzed (Participants) | 16 | 0 | 0 | 16
Age, Continuous [Mean (Full Range); unit: years] | 36 [21 to 70] |  |  | 36 [21 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 |  |  | 12
  Male | 4 |  |  | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 |  |  | 4
  Not Hispanic or Latino | 12 |  |  | 12
  Unknown or Not Reported | 0 |  |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 12 |  |  | 12
  Asian | 0 |  |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  |  | 0
  Black or African American | 0 |  |  | 0
  White | 3 |  |  | 3
  More than one race | 1 |  |  | 1
  Unknown or Not Reported | 0 |  |  | 0
Confidence communicating with Elders [Count of Participants; unit: Participants] — Qualitative self-report regarding confidence communicating with American Indian Elders about their health issues and healthcare and insurance options.
  Participants
    Comfortable communicating with AIEs about health and healthcare issues | 16 |  |  | 16
    Comfortable communicating with AIEs about health insurance | 11 |  |  | 11
    Uncomfortable communicating AIEs about insurance due to lack of knowledge | 3 |  |  | 3
    Experienced language barriers communicating with AIEs | 5 |  |  | 5
    Experienced challenges communicating with AIEs about difficult or taboo topics | 4 |  |  | 4
Confidence communicating with healthcare providers [Count of Participants; unit: Participants] — Qualitative self-report of confidence communicating with healthcare providers regarding the health needs, healthcare options, barriers to care, and insurance issues experienced by American Indian Elders.
  Participants
    Comfortable communicating with healthcare providers due to regular experience doing so | 12 |  |  | 12
    Comfortable communicating with healthcare providers when receiving referrals to help AIEs | 7 |  |  | 7
Comfort using Seasons of Care Guide [Count of Participants; unit: Participants] — Qualitative self-report of comfort using the Seasons of Care guide to help American Indian Elders as part of everyday work.
  Participants
    Comfortable using the Seasons of Care Guide in their work | 10 |  |  | 10
    Confident that they would become comfortable with the Seasons of Care Guide over time | 5 |  |  | 5
    Felt that the Seasons of Care Guide was no different than other resources they already used | 1 |  |  | 1

OUTCOME MEASURES:

1. Primary Outcome: User Evaluation Survey
Description: A semi-structured, in-person interview (or focus group, depending on availability) with AIEs and healthcare providers who interacted with a navigator using the Seasons of Care app to assess experiences with, and effects of, the Seasons of Care app; suggestions to improve the Seasons of Care app
Time Frame: Once at the end of P2 (Month 8 of 8)
Population: Due to the complete closure of tribal communities during the COVID-19 pandemic, no data were collected for this outcome measure.
Arm/Group | Navigators | American Indian Elders (AIEs) | Healthcare Providers/Staff
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Navigator Pre- and Post-Evaluation Interview
Description: A semi-structured, in-person interview comprised of open-ended questions to assess navigator's confidence and experiences with communicating health information to AIEs and healthcare providers; perceptions of the Seasons of Care app
Time Frame: Month 1 and 4 (of 8) for P1 Navigators; Month 5 and 8 (of 8) for P2 Navigators
Population: Due to the complete closure of tribal communities during the COVID-19 pandemic, focus groups with AIEs and healthcare providers/staff were not completed. Three Navigators were unable to complete post-evaluation interviews due to changing responsibilities during the COVID-19 pandemic. One Navigator left their position before completing the post-evaluation interview.
Measure: Count of Participants; unit: Participants
Arm/Group | Navigators | American Indian Elders (AIEs) | Healthcare Providers/Staff
Number analyzed (Participants) | 12 | 0 | 0
Participants
  Effects of Seasons of Care Guide on Communication with Providers: Improved | 3 |  |
  Effects of Seasons of Care Guide on Communication with Providers: Improved but with some remaining barriers | 2 |  |
  Effects of Seasons of Care Guide on Communication with Providers: No change | 1 |  |
  Effects of Seasons of Care Guide on Communication with Providers: No response | 6 |  |
  Effects of Seasons of Care Guide on Communication with Elders: Improved | 5 |  |
  Effects of Seasons of Care Guide on Communication with Elders: Improved but with some remaining barriers | 0 |  |
  Effects of Seasons of Care Guide on Communication with Elders: No change | 3 |  |
  Effects of Seasons of Care Guide on Communication with Elders: No response | 4 |  |

3. Other Pre Specified Outcome: User Evaluation Demographic Survey
Description: A demographic survey with AIEs and healthcare providers who interacted with a navigator using the Seasons of Care app
Time Frame: Once at the end of P2 (Month 8 of 8)
Population: Due to complete closure of tribal communities during the COVID-19 pandemic, no data were collected for this outcome measure.
Arm/Group | Navigators | American Indian Elders (AIEs) | Healthcare Providers/Staff
Number analyzed (Participants) | 0 | 0 | 0

4. Other Pre Specified Outcome: Feasibility Questionnaire
Description: A written questionnaire to assess navigator's experiences with, and effects of, Seasons of Care Guide
Time Frame: Assessed monthly for 4 months; participants' ratings for each category were averaged. Average ratings per participant for each category is reported here.
Population: Two Navigators were unable to complete any monthly questionnaires due to changing work responsibilities during the COVID-19 pandemic. One Navigator left their position before completing any questionnaires.
Measure: Count of Participants; unit: Participants
Arm/Group | Navigators | American Indian Elders (AIEs) | Healthcare Providers/Staff
Number analyzed (Participants) | 13 | 0 | 0
Participants
  Looks appealing (Average rating: 10=Strongly agree, 1=Strongly disagree): 10 | 4 |  |
  Looks appealing (Average rating: 10=Strongly agree, 1=Strongly disagree): 9 | 4 |  |
  Looks appealing (Average rating: 10=Strongly agree, 1=Strongly disagree): 8 | 3 |  |
  Looks appealing (Average rating: 10=Strongly agree, 1=Strongly disagree): 7 | 1 |  |
  Looks appealing (Average rating: 10=Strongly agree, 1=Strongly disagree): 6 | 0 |  |
  Looks appealing (Average rating: 10=Strongly agree, 1=Strongly disagree): 5 | 1 |  |
  Looks appealing (Average rating: 10=Strongly agree, 1=Strongly disagree): 4 | 0 |  |
  Looks appealing (Average rating: 10=Strongly agree, 1=Strongly disagree): 3 | 0 |  |
  Looks appealing (Average rating: 10=Strongly agree, 1=Strongly disagree): 2 | 0 |  |
  Looks appealing (Average rating: 10=Strongly agree, 1=Strongly disagree): 1 | 0 |  |
  Looks appealing (Average rating: 10=Strongly agree, 1=Strongly disagree): Not rated | 0 |  |
  Can easily navigate on first try (Average rating: 10=Strongly agree, 1=Strongly disagree): 10 | 3 |  |
  Can easily navigate on first try (Average rating: 10=Strongly agree, 1=Strongly disagree): 9 | 2 |  |
  Can easily navigate on first try (Average rating: 10=Strongly agree, 1=Strongly disagree): 8 | 6 |  |
  Can easily navigate on first try (Average rating: 10=Strongly agree, 1=Strongly disagree): 7 | 1 |  |
  Can easily navigate on first try (Average rating: 10=Strongly agree, 1=Strongly disagree): 6 | 0 |  |
  Can easily navigate on first try (Average rating: 10=Strongly agree, 1=Strongly disagree): 5 | 1 |  |
  Can easily navigate on first try (Average rating: 10=Strongly agree, 1=Strongly disagree): 4 | 0 |  |
  Can easily navigate on first try (Average rating: 10=Strongly agree, 1=Strongly disagree): 3 | 0 |  |
  Can easily navigate on first try (Average rating: 10=Strongly agree, 1=Strongly disagree): 2 | 0 |  |
  Can easily navigate on first try (Average rating: 10=Strongly agree, 1=Strongly disagree): 1 | 0 |  |
  Can easily navigate on first try (Average rating: 10=Strongly agree, 1=Strongly disagree): Not rated | 0 |  |
  Can easily re-located info (Average rating: 10=Strongly agree, 1=Strongly disagree): 10 | 3 |  |
  Can easily re-located info (Average rating: 10=Strongly agree, 1=Strongly disagree): 9 | 3 |  |
  Can easily re-located info (Average rating: 10=Strongly agree, 1=Strongly disagree): 8 | 5 |  |
  Can easily re-located info (Average rating: 10=Strongly agree, 1=Strongly disagree): 7 | 1 |  |
  Can easily re-located info (Average rating: 10=Strongly agree, 1=Strongly disagree): 6 | 0 |  |
  Can easily re-located info (Average rating: 10=Strongly agree, 1=Strongly disagree): 5 | 1 |  |
  Can easily re-located info (Average rating: 10=Strongly agree, 1=Strongly disagree): 4 | 0 |  |
  Can easily re-located info (Average rating: 10=Strongly agree, 1=Strongly disagree): 3 | 0 |  |
  Can easily re-located info (Average rating: 10=Strongly agree, 1=Strongly disagree): 2 | 0 |  |
  Can easily re-located info (Average rating: 10=Strongly agree, 1=Strongly disagree): 1 | 0 |  |
  Can easily re-located info (Average rating: 10=Strongly agree, 1=Strongly disagree): Not rated | 0 |  |
  Can find relevant info using "Search" (Average rating: 10=Strongly agree, 1=Strongly disagree): 10 | 5 |  |
  Can find relevant info using "Search" (Average rating: 10=Strongly agree, 1=Strongly disagree): 9 | 1 |  |
  Can find relevant info using "Search" (Average rating: 10=Strongly agree, 1=Strongly disagree): 8 | 6 |  |
  Can find relevant info using "Search" (Average rating: 10=Strongly agree, 1=Strongly disagree): 7 | 0 |  |
  Can find relevant info using "Search" (Average rating: 10=Strongly agree, 1=Strongly disagree): 6 | 0 |  |
  Can find relevant info using "Search" (Average rating: 10=Strongly agree, 1=Strongly disagree): 5 | 1 |  |
  Can find relevant info using "Search" (Average rating: 10=Strongly agree, 1=Strongly disagree): 4 | 0 |  |
  Can find relevant info using "Search" (Average rating: 10=Strongly agree, 1=Strongly disagree): 3 | 0 |  |
  Can find relevant info using "Search" (Average rating: 10=Strongly agree, 1=Strongly disagree): 2 | 0 |  |
  Can find relevant info using "Search" (Average rating: 10=Strongly agree, 1=Strongly disagree): 1 | 0 |  |
  Can find relevant info using "Search" (Average rating: 10=Strongly agree, 1=Strongly disagree): Not rated | 0 |  |
  Can easily find healthcare facilities (Average rating: 10=Strongly agree, 1=Strongly disagree): 10 | 1 |  |
  Can easily find healthcare facilities (Average rating: 10=Strongly agree, 1=Strongly disagree): 9 | 5 |  |
  Can easily find healthcare facilities (Average rating: 10=Strongly agree, 1=Strongly disagree): 8 | 3 |  |
  Can easily find healthcare facilities (Average rating: 10=Strongly agree, 1=Strongly disagree): 7 | 2 |  |
  Can easily find healthcare facilities (Average rating: 10=Strongly agree, 1=Strongly disagree): 6 | 2 |  |
  Can easily find healthcare facilities (Average rating: 10=Strongly agree, 1=Strongly disagree): 5 | 0 |  |
  Can easily find healthcare facilities (Average rating: 10=Strongly agree, 1=Strongly disagree): 4 | 0 |  |
  Can easily find healthcare facilities (Average rating: 10=Strongly agree, 1=Strongly disagree): 3 | 0 |  |
  Can easily find healthcare facilities (Average rating: 10=Strongly agree, 1=Strongly disagree): 2 | 0 |  |
  Can easily find healthcare facilities (Average rating: 10=Strongly agree, 1=Strongly disagree): 1 | 0 |  |
  Can easily find healthcare facilities (Average rating: 10=Strongly agree, 1=Strongly disagree): Not rated | 0 |  |
  AIEs like using it (Average rating: 10=Strongly agree, 1=Strongly disagree): 10 | 1 |  |
  AIEs like using it (Average rating: 10=Strongly agree, 1=Strongly disagree): 9 | 2 |  |
  AIEs like using it (Average rating: 10=Strongly agree, 1=Strongly disagree): 8 | 3 |  |
  AIEs like using it (Average rating: 10=Strongly agree, 1=Strongly disagree): 7 | 1 |  |
  AIEs like using it (Average rating: 10=Strongly agree, 1=Strongly disagree): 6 | 1 |  |
  AIEs like using it (Average rating: 10=Strongly agree, 1=Strongly disagree): 5 | 1 |  |
  AIEs like using it (Average rating: 10=Strongly agree, 1=Strongly disagree): 4 | 1 |  |
  AIEs like using it (Average rating: 10=Strongly agree, 1=Strongly disagree): 3 | 2 |  |
  AIEs like using it (Average rating: 10=Strongly agree, 1=Strongly disagree): 2 | 1 |  |
  AIEs like using it (Average rating: 10=Strongly agree, 1=Strongly disagree): 1 | 0 |  |
  AIEs like using it (Average rating: 10=Strongly agree, 1=Strongly disagree): Not rated | 0 |  |
  Useful for working with AIEs: 10 | 3 |  |
  Useful for working with AIEs: 9 | 3 |  |
  Useful for working with AIEs: 8 | 2 |  |
  Useful for working with AIEs: 7 | 2 |  |
  Useful for working with AIEs: 6 | 1 |  |
  Useful for working with AIEs: 5 | 1 |  |
  Useful for working with AIEs: 4 | 1 |  |
  Useful for working with AIEs: 3 | 0 |  |
  Useful for working with AIEs: 2 | 0 |  |
  Useful for working with AIEs: 1 | 0 |  |
  Useful for working with AIEs: Not rated | 0 |  |
  Provides info not available elsewhere (Average rating: 10=Strongly agree, 1=Strongly disagree): 10 | 2 |  |
  Provides info not available elsewhere (Average rating: 10=Strongly agree, 1=Strongly disagree): 9 | 0 |  |
  Provides info not available elsewhere (Average rating: 10=Strongly agree, 1=Strongly disagree): 8 | 5 |  |
  Provides info not available elsewhere (Average rating: 10=Strongly agree, 1=Strongly disagree): 7 | 2 |  |
  Provides info not available elsewhere (Average rating: 10=Strongly agree, 1=Strongly disagree): 6 | 2 |  |
  Provides info not available elsewhere (Average rating: 10=Strongly agree, 1=Strongly disagree): 5 | 2 |  |
  Provides info not available elsewhere (Average rating: 10=Strongly agree, 1=Strongly disagree): 4 | 0 |  |
  Provides info not available elsewhere (Average rating: 10=Strongly agree, 1=Strongly disagree): 3 | 0 |  |
  Provides info not available elsewhere (Average rating: 10=Strongly agree, 1=Strongly disagree): 2 | 0 |  |
  Provides info not available elsewhere (Average rating: 10=Strongly agree, 1=Strongly disagree): 1 | 0 |  |
  Provides info not available elsewhere (Average rating: 10=Strongly agree, 1=Strongly disagree): Not rated | 0 |  |
  Useful tool for healthcare providers (Average rating: 10=Strongly agree, 1=Strongly disagree): 10 | 2 |  |
  Useful tool for healthcare providers (Average rating: 10=Strongly agree, 1=Strongly disagree): 9 | 1 |  |
  Useful tool for healthcare providers (Average rating: 10=Strongly agree, 1=Strongly disagree): 8 | 6 |  |
  Useful tool for healthcare providers (Average rating: 10=Strongly agree, 1=Strongly disagree): 7 | 2 |  |
  Useful tool for healthcare providers (Average rating: 10=Strongly agree, 1=Strongly disagree): 6 | 0 |  |
  Useful tool for healthcare providers (Average rating: 10=Strongly agree, 1=Strongly disagree): 5 | 2 |  |
  Useful tool for healthcare providers (Average rating: 10=Strongly agree, 1=Strongly disagree): 4 | 0 |  |
  Useful tool for healthcare providers (Average rating: 10=Strongly agree, 1=Strongly disagree): 3 | 0 |  |
  Useful tool for healthcare providers (Average rating: 10=Strongly agree, 1=Strongly disagree): 2 | 0 |  |
  Useful tool for healthcare providers (Average rating: 10=Strongly agree, 1=Strongly disagree): 1 | 0 |  |
  Useful tool for healthcare providers (Average rating: 10=Strongly agree, 1=Strongly disagree): Not rated | 0 |  |
  Is helping AIEs access care and insurance (Average rating: 10=Strongly agree, 1=Strongly disagree): 10 | 2 |  |
  Is helping AIEs access care and insurance (Average rating: 10=Strongly agree, 1=Strongly disagree): 9 | 2 |  |
  Is helping AIEs access care and insurance (Average rating: 10=Strongly agree, 1=Strongly disagree): 8 | 4 |  |
  Is helping AIEs access care and insurance (Average rating: 10=Strongly agree, 1=Strongly disagree): 7 | 0 |  |
  Is helping AIEs access care and insurance (Average rating: 10=Strongly agree, 1=Strongly disagree): 6 | 0 |  |
  Is helping AIEs access care and insurance (Average rating: 10=Strongly agree, 1=Strongly disagree): 5 | 1 |  |
  Is helping AIEs access care and insurance (Average rating: 10=Strongly agree, 1=Strongly disagree): 4 | 3 |  |
  Is helping AIEs access care and insurance (Average rating: 10=Strongly agree, 1=Strongly disagree): 3 | 0 |  |
  Is helping AIEs access care and insurance (Average rating: 10=Strongly agree, 1=Strongly disagree): 2 | 0 |  |
  Is helping AIEs access care and insurance (Average rating: 10=Strongly agree, 1=Strongly disagree): 1 | 0 |  |
  Is helping AIEs access care and insurance (Average rating: 10=Strongly agree, 1=Strongly disagree): Not rated | 1 |  |

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from Navigators monthly during Phase 1 and Phase 2
Description: Due to the complete closure of tribal communities during the COVID-19 pandemic, focus groups with AIEs and healthcare providers were not completed
Arm/Group | Navigators | American Indian Elders (AIEs) | Healthcare Providers/Staff
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/16 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Data collection with American Indian Elders and healthcare providers/staff to evaluate their experiences with the Seasons of Care Guide was not possible due to the closure of tribal communities during the COVID-19 pandemic and the infeasibility of collecting data with these participants remotely. These evaluation data are qualitative; future research on the dissemination of the Seasons of Care Guide should prioritize quantitative methods.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-07): https://cdn.clinicaltrials.gov/large-docs/04/NCT03550404/Prot_SAP_000.pdf
  • Informed Consent Form (2016-09-15): https://cdn.clinicaltrials.gov/large-docs/04/NCT03550404/ICF_001.pdf